CLINICAL TRIAL: NCT01376726
Title: A Phase I Open-Label Trial to Evaluate the Safety and Immunogenicity of an HIV-1 Subtype C gp140 Vaccine With MF59 Adjuvant in Healthy, HIV-1 Uninfected Adult Participants Previously Primed or Unprimed With HIV-1 Subtype B Envelope Subunit Vaccines With MF59
Brief Title: Evaluating the Safety and Immune Response to an HIV Vaccine in Healthy, HIV-Uninfected Adults Who Have Participated in Previous HIV Vaccine Clinical Trials and in Adults Who Have Not Participated in Previous HIV Vaccine Clinical Trials
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Novartis Vaccines and Diagnostics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 088; 11779 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Previous HIV Vaccine Trial Participants (Group 1) (Experimental): Participants will receive the study vaccine administered as one 0.5 mL intramuscular injection (IM) in either deltoid at baseline and Month 6.
  Participants in the study extension will receive an additional injection of the study vaccine approximately 14 to 20 months after their second (Month 6) vaccination.
  Interventions: Biological: Sub C gp140 Vaccine; Biological: MF59C.1 Adjuvant
- No Previous HIV Vaccine Trial (Group 2) (Experimental): Participants will receive the study vaccine administered as one 0.5 mL IM in either deltoid at baseline and Month 6.
  Participants in the study extension will receive an additional injection of the study vaccine approximately 14 to 20 months after their second (Month 6) vaccination.
  Interventions: Biological: Sub C gp140 Vaccine; Biological: MF59C.1 Adjuvant

INTERVENTIONS:
Biological: Sub C gp140 Vaccine — Sub C gp140 100 mcg will be combined with MF59C.1 and administered as one injection (0.5 mL) IM in either deltoid at baseline and Month 6.
  Participants in the study extension will receive an additional injection of the study vaccine approximately 14 to 20 months after their second (Month 6) vaccination.
Biological: MF59C.1 Adjuvant — Sub C gp140 100 mcg will be combined with MF59C.1 and administered as one injection (0.5 mL) IM in either deltoid at baseline and Month 6.
  Participants in the study extension will receive an additional injection of the study vaccine approximately 14 to 20 months after their second (Month 6) vaccination.

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to an HIV vaccine in healthy, HIV-uninfected adults who have participated in a previous HIV vaccine clinical trial and in healthy, HIV-uninfected adults who have not participated in a previous HIV vaccine clinical trial.

DETAILED DESCRIPTION:
Previous clinical trials have shown that people who receive a second vaccine for certain conditions after having received a prior vaccine may have a better antibody response to the second vaccine than people who receive the vaccine for the first time. This is known as "priming" and it may occur in people receiving a second vaccine even if the first vaccine was received several years previously. This study will enroll healthy, HIV-uninfected adults who have participated in a previous HIV vaccine clinical trial and received HIV-1 subtype B envelope subunit vaccines with MF59 adjuvant, and healthy, HIV-uninfected adults who have not participated in a previous HIV vaccine clinical trial and therefore have not previously received any HIV vaccines. Participants in this study will receive a total of two injections, each 6 months apart, of the HIV-1 Sub Cgp140 vaccine with MF59 adjuvant. Researchers will evaluate the safety and immune response to the study vaccine and determine if people who participated in a previous HIV vaccine clinical trial demonstrate an improved antibody response to the study vaccine versus people who have never received an HIV vaccine.

This study will enroll two groups of participants. Group 1 will include healthy, HIV-uninfected adults who have participated in a previous HIV vaccine clinical trial. Group 2 will include healthy, HIV-uninfected adults who have not participated in an HIV vaccine clinical trial. All participants will receive the study vaccine injected into their upper arm at baseline and Month 6.

At the baseline study visit, all participants will undergo a physical examination, a medical and medication history review, and blood collection. Female participants will also take a pregnancy test. Participants will complete questionnaires and receive counseling on HIV risk reduction and pregnancy prevention. Saliva samples will be obtained from all participants and rectal fluids, semen samples, and cervical secretions will be obtained from some participants. After receiving the vaccine, participants will remain in the clinic for at least 30 minutes for observation and monitoring of side effects. For 3 days after the vaccination, participants will record any side effects in a symptom log.

Participants in Group 1 will attend study visits 1 and 2 weeks after the first vaccination study visit, at Month 6 for the second vaccination, 1 and 2 weeks after the Month 6 study visit, and at Months 9 and 12. Participants in Group 2 will attend study visits 1 and 3 days and 1 and 2 weeks after the first vaccination study visit, at Month 6 for the second vaccination, 1 and 3 days and 1 and 2 weeks after the Month 6 study visit, and at Months 9 and 12. Follow-up study visits will include select study procedures. Blood collected during study visits may be saved for future testing. Study researchers will contact participants at Month 18 for follow-up health monitoring.

In July 2013, an extension to the study was announced. Current study participants will be screened to see if they are eligible to participate in the study extension. Participants who are eligible will receive one additional injection of the study vaccine, at a visit approximately 14 to 20 months after their second (Month 6) vaccination. Additional study visits will occur 2 weeks, and 3 and 6 months after receiving the third vaccination. Select visits will include a physical examination, blood collection, saliva collection, pregnancy test for female participants, HIV testing and risk reduction counseling, and interviews and questionnaires. Study researchers will contact participants 1 year after the third vaccination for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HVTN Clinical Research Site (CRS) and willing to be followed for the planned duration of the study
* Able and willing to provide informed consent
* Assessment of understanding: must demonstrate understanding of this study and the Step Study results; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to receive HIV test results
* Willing to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required study clinic visit
* Assessed by the clinic staff as being at low risk for HIV infection
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required study clinic visit
* In good general health as shown by medical history, physical exam, and screening laboratory tests
* For Group 1: Prior receipt of an HIV-1 subtype B envelope subunit vaccine (gp120, gp140) with MF59 adjuvant. More information on this criterion can be found in the protocol.
* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female, greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell (WBC) count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3
* Chemistry panel: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 1.25 times the upper limit of normal; creatinine less than or equal to the institutional upper limits of normal
* Negative HIV-1 and -2 blood test: Group 1 (primed) participants must have a negative test result for HIV infection following the HVTN Lab Program's in-study HIV testing algorithm. Group 2 (unprimed) participants must have a negative test result for HIV-infection following the CRS's routine HIV screening procedures with an FDA-approved blood test.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine: Negative urine glucose, negative or trace urine protein, and negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis within institutional normal range)
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Participants who were born female must agree to consistently use effective contraception from at least 21 days prior to enrollment through the last required protocol clinic visit for sexual activity that could lead to pregnancy, or not be of reproductive potential, or be sexually abstinent. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization, until after the last required study clinic visit
* Participants who were born female and agree to cervical fluid collection must report having a normal Pap smear or atypical squamous cells of undetermined significance (ASCUS) with no evidence of high risk HPV within 3 years prior to enrollment in order to participate in cervical mucosal sampling. This is not a requirement for study entry.

Inclusion Criteria for Study Extension:

Prior to participation in the study extension, participants will be rescreened for eligibility. The participant must have received the two earlier vaccinations in the study.

Participants must demonstrate understanding of the study extension and complete a questionnaire prior to receiving the third vaccination; however, understanding of the Step study results will not be specifically reassessed.

Study extension participants must have a negative test result for HIV infection following the HVTN Lab Program's in-study HIV testing algorithm, within 21 days prior to receipt of the third vaccination.

All inclusion criteria listed above for the study still apply EXCEPT the following criteria:

* Age of 18 to 55 years
* Assessment of understanding
* Prior receipt of an HIV-1 subtype B envelope subunit vaccine (gp120, gp140) with MF59 adjuvant (Group 1 participants)
* Negative hepatitis B surface antigen (HBsAg), and negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive. Repeat testing is not necessary for syphilis and hepatitis B and C, which will be excluded based on updated participant medical history.
* Normal Pap smear or atypical squamous cells of undetermined significance (ASCUS) criteria with no evidence of high risk HPV within 3 years prior to enrollment in order to participate in cervical mucosal sampling.

Exclusion Criteria:

* History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B within the 12 months prior to study entry
* Untreated or incompletely treated syphilis infection
* For Group 2 only: HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, the HVTN 088 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) or adjuvant(s) other than MF59 received within the 5 years prior to study entry in a prior vaccine trial. Exceptions may be made for vaccines/adjuvants that have subsequently undergone licensure by the FDA. For potential participants who have received an experimental vaccine(s)/adjuvant(s) greater than 5 years before study entry, eligibility for enrollment will be determined by the PSRT on a case-by-case basis. For potential participants who have received control/placebo in an experimental vaccine trial, the HVTN 088 PSRT will determine eligibility on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines (e.g., pneumococcal, tetanus, hepatitis A or B) and were received within 14 days prior to any vaccination
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to study entry].)
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the study
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, study adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the 12 months before study entry
* History of hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Hypertension: If a person has been diagnosed with hypertension during screening or previously, exclude for hypertension that is not well controlled. If a person has NOT been diagnosed with hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at study entry or diastolic blood pressure greater than or equal to 100 mm Hg at study entry. More information on this criterion can be found in the protocol.
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with two or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, platelet disorder requiring special precautions)
* Cancer (Not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.)
* Seizure disorder (Not excluded: a participant with a history of seizures who has not required medications or had a seizure within the 3 years prior to study entry.)
* Asplenia: any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the study. Specifically excluded are people with psychoses within the 3 years prior to study entry, ongoing risk for suicide, or history of suicide attempt or gesture within the 3 years prior to study entry.
* Pregnant or breastfeeding

Exclusion Criteria for Optional Mucosal Sampling:

* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to the planned procedure

Exclusion Criteria for Study Extension:

Prior to participation in the study extension, participants will be rescreened for eligibility. The participant must have received the two earlier vaccinations in the study. All exclusion criteria listed above for the study still apply EXCEPT the following criteria:

* HIV vaccine(s) received in a prior HIV vaccine trial (Group 2 participants)
* BMI greater than or equal to 40; or BMI greater than or equal to 35 with two or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Frequency of severe local and systemic reactogenicity signs and symptoms | Measured within the first 3 days after vaccination
Summary reports of the frequency of adverse events (AEs) by group, by body system, MedDRA preferred term, severity, and assessed relationship to study product | Measured through 12 months post last vaccination
All serious adverse events (SAEs) | Measured through 12 months post last vaccination
Laboratory measures of safety at baseline and following vaccinations: descriptive analyses of white blood cells (WBC), neutrophils, lymphocytes, hemoglobin, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatinine | Measured through 3 months post last vaccination
Neutralizing antibody titers to SF162 and TV1 | Measured through 6 months post last vaccination
Neutralizing antibody titers and breadth against heterologous primary isolates | Measured through 6 months post last vaccination

SECONDARY OUTCOMES:
SF162 Env-specific non-neutralizing antibodies and TV1 Env-specific antibodies as determined by multiplex antibody assays | Measured through 6 months post last vaccination
ConS gp140 specific IgG subclass characterization (IgG1- IgG4) and IgA measurement by custom HIV-1 multiplex assay | Measured through 6 months post last vaccination
Intracellular cytokine staining to evaluate polyfunctional cytokine responses by antigen-specific CD4 T cells | Measured through 6 months post last vaccination
Lymphoproliferation of antigen-specific CD4 T cells by carboxyfluorescein diacetate succinimidyl ester (CFSE) assay | Measured through 6 months post last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Paul Spearman, Study Chair — Emory University
Locations (3):
- United States (3):
  - Alabama CRS, Birmingham, Alabama
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Background] Goepfert PA, Tomaras GD, Horton H, Montefiori D, Ferrari G, Deers M, Voss G, Koutsoukos M, Pedneault L, Vandepapeliere P, McElrath MJ, Spearman P, Fuchs JD, Koblin BA, Blattner WA, Frey S, Baden LR, Harro C, Evans T; NIAID HIV Vaccine Trials Network. Durable HIV-1 antibody and T-cell responses elicited by an adjuvanted multi-protein recombinant vaccine in uninfected human volunteers. Vaccine. 2007 Jan 5;25(3):510-8. doi: 10.1016/j.vaccine.2006.07.050. Epub 2006 Aug 10. PMID 17049679
- [Background] Scheid JF, Mouquet H, Feldhahn N, Seaman MS, Velinzon K, Pietzsch J, Ott RG, Anthony RM, Zebroski H, Hurley A, Phogat A, Chakrabarti B, Li Y, Connors M, Pereyra F, Walker BD, Wardemann H, Ho D, Wyatt RT, Mascola JR, Ravetch JV, Nussenzweig MC. Broad diversity of neutralizing antibodies isolated from memory B cells in HIV-infected individuals. Nature. 2009 Apr 2;458(7238):636-40. doi: 10.1038/nature07930. Epub 2009 Mar 15. PMID 19287373